CLINICAL TRIAL: NCT07228754
Title: How Realistic Are Caregivers' Expectations in Determining Rehabilitation Goals for Subacute Stroke Patients?
Brief Title: How Realistic Are Caregivers' Expectations in Patients With Subacute Stroke?
Status: Recruiting | Type: Observational
Sponsor: Ankara Etlik City Hospital (Other Government)
Responsible Party: Principal Investigator, Ayse Naz Kalem, PM&R Specialist, Ankara Etlik City Hospital
Other Study IDs: AEŞH-BADEK1-2025-479
Record Dates: First submitted 2025-11-13; First posted 2025-11-14 (Actual); Last update posted 2025-11-14 (Actual); Status verified 2025-11

CONDITIONS: Stroke Rehabilitation; Stroke Rehabilitation and Caregivers

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Stoke Patients
  Interventions: Other: Conventional rehabilitation programme

INTERVENTIONS:
Other: Conventional rehabilitation programme — Conventional rehabilitation programme described for patients individually

SUMMARY:
The aim of this study is to evaluate the extent to which the patient's goals and the physical therapist's goals can be achieved after stroke rehabilitation and to compare their expectations in terms of rehabilitation outcomes. Thus, the expected benefit of the study is to contribute to goal setting in post-stroke rehabilitation. There are no expected risks from the study.

ELIGIBILITY:
Inclusion Criteria:

1. Followed by ischemic or hemorrhagic stroke
2. No more than 6 months have passed since the date of the event
3. Being between the ages of 18 and 75
4. The caregiver being between the ages of 18 and 75

Exclusion Criteria:

1. The patient has additional neurological conditions besides stroke
2. The patient has a psychiatric condition
3. The patient is not willing to participate in the study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Fifty-eight stroke patients receiving inpatient treatment at the Ankara Etlik City Hospital Brain Injury-3 clinic and their caregivers will be evaluated.
Sampling Method: Probability Sample
Enrollment: 58 (Estimated)
Dates: Start 2025-11-06 (Actual); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
Goal Attainment Scale | First day of rehabilitation, 4th week of rehabilitation
  The Goal Attainment Scale will be used as the primary outcome measure within the framework of goals set separately by the caregiver and the physical therapist.

SECONDARY OUTCOMES:
Functional Ambulation Scale | First day of rehabilitation, 4th week of rehabilitation
Modified Barthel Index | First day of rehabilitation, 4th week of rehabilitation

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara Etlik City Hospital, Ankara, Yenimahalle, Turkey (Türkiye)